CLINICAL TRIAL: NCT02154048
Title: Analgesic Efficacy of Perineural Dexamethasone Added to Ropivacaine 0.5% With 1:400,000 Epinephrine During Single-injection Supraclavicular Block for Outpatient Hand Surgery
Brief Title: Analgesic Efficacy of Perineural Dexamethasone During Supraclavicular Block for Hand Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00019301
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Surgery, Hand
MeSH Terms: interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ropivacaine + dexamethasone (Active Comparator): This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with 1:400,000 epinephrine and an IV preservative-free dexamethasone 8 mg injection.
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone
- ropivacaine + placebo (Placebo Comparator): This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with 1:400,000 epinephrine and an intravenous (IV) normal saline placebo injection.
  Interventions: Drug: Ropivacaine; Other: Placebo
- ropivacaine + dexamethasone + placebo (Active Comparator): This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with both 1:400,000 epinephrine and preservative-free dexamethasone 8mg and an IV normal saline placebo injection.
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone; Other: Placebo

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Naropin
Drug: Dexamethasone
  Arms: ropivacaine + dexamethasone; ropivacaine + dexamethasone + placebo
Other: Placebo
  Arms: ropivacaine + dexamethasone + placebo; ropivacaine + placebo

SUMMARY:
The purpose of this study is to determine whether the addition of dexamethasone prolongs analgesia when added to long-acting local anesthetic during single-injection supraclavicular block for outpatient hand surgery.

DETAILED DESCRIPTION:
The goal for pain control after surgery is to provide the best possible pain control for the longest period of time with the least amount of side effects. One type of pain medication is called local anesthetic, which is a numbing medication that is injected in the area surrounding nerves to block pain. This injection is called a nerve block. Ropivacaine is a local anesthetic that is commonly used for nerve blocks and will be used in this study. The effects of ropivacaine may last for 8 to 12 hours after surgery. Recent research studies have shown that adding a medication called dexamethasone (a steroid) may increase the time that the nerve block will provide pain control. The purpose of this study is to see if adding dexamethasone to ropivacaine and injecting this around the nerves during a supraclavicular brachial plexus block increases the duration of pain relief as compared to both placebo control and systemic control groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients scheduled for elective outpatient hand surgery with same day discharge at the Duke Ambulatory Surgery Center

Exclusion Criteria:

* Patients who refuse regional anesthesia
* Patients in whom peripheral nerve block is contraindicated
* Patients unable to sign/understand consent
* Patients with significant language barriers who cannot comply with data collection process
* Patients with known allergies to local anesthetics
* Pregnancy
* Chronic pain patients or patients requiring chronic opioid treatment
* Patients with a history of diabetes
* Patients with contraindication to steroid administration (allergy, chronic steroid use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Melton, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because the required sample size of 60 subjects was not met, the study was terminated. Five subjects were enrolled from April 2012 to September 2013.
Groups:
- Intravenous (IV) Control Group: This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with 1:400,000 epinephrine and an IV preservative-free dexamethasone 8 mg injection.
  Ropivacaine + Dexamethasone
- Local Anesthetic (LA) Control Group: This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with 1:400,000 epinephrine and an intravenous (IV) normal saline placebo injection.
  Ropivacaine + Placebo
- Additive Group: This group will be comprised of 20 subjects who will receive an ultrasound-guided supraclavicular brachial plexus block with 30ml of ropivacaine 0.5% with both 1:400,000 epinephrine and preservative-free dexamethasone 8mg and an IV normal saline placebo injection.
  Ropivacaine + Dexamethasone + Placebo
Period: Overall Study
Arm/Group | Intravenous (IV) Control Group | Local Anesthetic (LA) Control Group | Additive Group
Started | 2 | 2 | 1
Completed | 2 | 2 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous (IV) Control Group | Local Anesthetic (LA) Control Group | Additive Group | Total
Number analyzed (Participants) | 2 | 2 | 1 | 5
Age, Customized [Number; unit: participants]
  >= 18 years | 2 | 2 | 1 | 5
  <=17 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 1 | 0 | 1 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Analgesic Dose
Time Frame: 48 hours
Population: one subject in the Local Anesthetic (LA) Control Group was not analyzed because subject did not return the data sheet
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Local Anesthetic (LA) Control Group | Intravenous (IV) Control Group | Additive Group
Number analyzed (Participants) | 1 | 2 | 1
hours | 10 (0) | 6 (0) | 4 (0)

ADVERSE EVENTS:
Arm/Group | Intravenous (IV) Control Group | Local Anesthetic (LA) Control Group | Additive Group
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No